CLINICAL TRIAL: NCT03140800
Title: Intrauterine Contraceptive Device:Clinical and Sonographic Correlation in Patients Presenting With Bleeding
Brief Title: Use Sonography in Patients With Intrauterine Device Presenting With Bleeding
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ESShafeek, Dr, Assiut University
Other Study IDs: IUD
Record Dates: First submitted 2017-05-03; First posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Contraception
MeSH Terms: interventions — Intrauterine Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intrauterine device — a method of contraception inserted in the uterus

SUMMARY:
Intrauterine contraceptive device is one of the most efficient and reversible methods of birth control with low cost and long duration of use However, in the first year after insertion, between 5 and 15% of women will have their Intrauterine contraceptive device removed because of irregular uterine bleeding which have been attributed to the effect of contact between the device and the endometrium and even the pressure on the uterine muscle . The disharmonious relationship between the Intrauterine contraceptive device and the uterus is the cause of most of the bleeding complaints, so bleeding is related to improper position rather than the contraceptive method itself which should be excluded before abandoning the Intrauterine contraceptive device for any other method of birth control

ELIGIBILITY:
Inclusion Criteria:

patients using intrauterine contraceptive device complaining of bleeding

Exclusion Criteria:

* a-Associated uterine, cervical,or adenexal pathology b-Associated pelvic infection c-Generalized bleeding disorders d-Medications causing coagulation defects e-Medical disorders causing bleeding e.g hypertention f-Endocrine disorder as thyroid dysfunction g-Who refuse to share in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients using intrauterine contraceptive device complaining of bleeding
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The intrauterine device-Endometrial distance | 3 months

IPD SHARING:
Plan to Share IPD: No